CLINICAL TRIAL: NCT01260402
Title: Randomized Comparison of Endocardial Versus Epicardial - From the Coronary Sinus - Left Ventricular Pacing for Resynchronization in Heart Failure.
Acronym: EPI-ENDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2010/12
Record Dates: First submitted 2010-12-08; First posted 2010-12-15 (Estimated); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Heart Failure; Cardiomyopathy, Dilated; Coronary Disease
Keywords: heart failure; Cardiomyopathy, dilated; Coronary disease; Cardiac Pacing, Artificial; cardiac resynchronization therapy; Hemodynamics; Randomized Controlled Trials; Open Study
MeSH Terms: conditions — Heart Failure; Cardiomyopathy, Dilated; Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epicardial (Active Comparator)
  Interventions: Device: Resynchronization using a coronary sinus approach
- Endocardial (Experimental)
  Interventions: Device: Resynchronization using a transeptal approach

INTERVENTIONS:
Device: Resynchronization using a transeptal approach — Cardiac resynchronization with one in the right ventricle and one in the left ventricle via a transeptal puncture.
  Devices used for procedure : Medtronic C304 or 6227DEF, Nykanen RF Wire, RADI PressureWire
  Arms: Endocardial
Device: Resynchronization using a coronary sinus approach — Cardiac resynchronization with one in the right ventricle and one in the left ventricle via the coronary sinus.
  Devices used for procedure : RADI PressureWire, routine catheters chosen by operator
  Arms: Epicardial

SUMMARY:
Biventricular pacing is a validated treatment for patients suffering from heart failure resistant to medical treatment. However, up to 30% of the patients are non responsive to this strategy using the coronary sinus approach to pace the Left Ventricle (LV).

It has been demonstrated that the magnitude of the improvement was highly dependant on the LV pacing site. The coronary sinus approach rarely offers more than 1 or 2 potential pacing sites. Resynchronisation using a transeptal approach to pace the left ventricle on the cardiology has been shown feasible on small series. We therefore would like to compare these two approached in a randomised prospective study to confirm the hypotheses that endocardial LV pacing by offering multiple choices for the pacing sites reduces the number of non responders and is associated with greater hemodynamic benefit when compared to the conventional coronary sinus approach.

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged 18 or above)
* Cardiac insufficiency of whatever cause (ischemic or non-ischemic)
* Left ventricular ejection fraction <35%
* NYHA Class III or IV with optimal medical treatment
* QRS duration > 120 ms
* Sinus rhythm
* Patient must have signed informed consent
* Patient must be registered in the national health care system

Exclusion Criteria:

* Aged under 18
* Patient with a mitral or aortic prosthesis
* Patient with contraindication to anti-coagulants
* Pregnant women
* Participation in another study
* Patient with contraindication for left ventricle catheterization by retrograde aortic approach , as a severe aortic stenosis requiring surgery, or an ascending aorta aneurism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-03-03 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-07-30 (Actual)

PRIMARY OUTCOMES:
the acute hemodynamic response judged by dP/dt max | Visit 3 : implantation day, during pacing procedure
  The primary outcome will be the acute hemodynamic response of the randomized pacing modality (endocardial vs epicardial Left Ventricle pacing) as judged by the highest gain in dP/dt max

SECONDARY OUTCOMES:
Implant success rate | Visit 3 : implantation day, end of pacing procedure
number of left ventricular pacing sites assessed | Visit 3 : implantation day, end of pacing procedure
Pacing Procedure duration | Visit 3 : implantation day, end of pacing procedure
Per and post implantation complications rate | Visit 4 : within 7 days after pacing procedure
Post implantation echocardiography comparing spontaneous rhythm and biventricular pacing for left ventricle ejection fraction | within 7 days after pacing procedure
Post implantation echocardiography comparing spontaneous rhythm and biventricular pacing for mitral regurgitation | within 7 days after pacing procedure
Post implantation echocardiography comparing spontaneous rhythm and biventricular pacing for atrioventricular asynchronism | within 7 days after pacing procedure
Post implantation echocardiography comparing spontaneous rhythm and biventricular pacing for inter and intra-ventricular asynchronism | within 7 days after pacing procedure
sensing performances of left ventricle pacing leads | within 7 days after pacing procedure
pacing threshold performances of left ventricle pacing leads | within 7 days after pacing procedure
impedances performances of left ventricle pacing leads | within 7 days after pacing procedure
Complications rate at 6 month Follow up | Visit 6 : 6-months after pacing procedure
Clinical benefit at 6 month Follow up: Gain in NYHA | 6-months after pacing procedure
Clinical benefit at 6 month Follow up: 6 minutes walk test | 6-months after pacing procedure
Clinical benefit at 6 month Follow up: quality of life questionnaire as compared to pre implantation | 6-months after pacing procedure
Echocardiography at 6 month Follow up: as compared to pre implantation for Left Ventricular Ejection Fraction | 6-months after pacing procedure
Echocardiography at 6 month Follow up: as compared to pre implantation for Left Ventricle volumes | 6-months after pacing procedure
Echocardiography at 6 month Follow up: as compared to pre implantation for mitral regurgitation | 6-months after pacing procedure
Echocardiography at 6 month Follow up: as compared to pre implantation for atrioventricular asynchronism | 6-months after pacing procedure
Echocardiography at 6 month Follow up: as compared to pre implantation for inter and intra-ventricular asynchronism | 6-months after pacing procedure
sensing performances of Left Ventricle pacing leads at 6 month Follow up | 6-months after pacing procedure
pacing threshold performances of Left Ventricle pacing leads at 6 month Follow up | 6-months after pacing procedure
impedances performances of Left Ventricle pacing leads at 6 month Follow up | 6-months after pacing procedure

CONTACTS AND LOCATIONS:
Overall Officials: Pierre JAIS, MD, Principal Investigator — University Hospital Bordeaux, France
Locations (1):
- Cardiologic Hospital Haut l'évêque, Pessac, France